CLINICAL TRIAL: NCT01398475
Title: Relative Bioavailability of the LY3009104 Free Base Test Formulation Compared to the Reference Phosphate Salt Formulation and the Effect of Food on the Bioavailability of the Test Formulation in Healthy Subjects
Brief Title: A Relative Bioavailability and Food Effect Study of New Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14016; I4V-MC-JADH (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Chronic Inflammatory Disorder; Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY3009104 Reference Formulation (Experimental): 8 milligrams (mg) LY3009104 (two 4-mg phosphate salt capsules), administered orally in the fasted state, once only. There will be a washout period of 5 to 7 days between doses of study drug.
  Interventions: Drug: LY3009104
- LY3009104 Test Formulation 1 (Experimental): 8 mg LY3009104 (one 8-mg smaller particle free base tablet), administered orally in the fasted state, once only. There will be a washout period of 5 to 7 days between doses of study drug.
  Interventions: Drug: LY3009104
- LY3009104 Test Formulation 2 (Experimental): 8 mg LY3009104 (one 8-mg larger particle free base tablet), administered orally in the fasted state, once only. There will be a washout period of 5 to 7 days between doses of study drug.
  Interventions: Drug: LY3009104
- LY3009104 Test Formulation 2 + Meal (Experimental): 8 mg LY3009104 (one 8-mg larger particle free base tablet), administered orally with high-fat/high calorie meal, once only. There will be a washout period of 5 to 7 days between doses of study drug.
  Interventions: Drug: LY3009104

INTERVENTIONS:
Drug: LY3009104 — Administered orally

SUMMARY:
The purpose of this trial is to assess the effect of 3 formulations on the relative bioavailability of LY3009104. Participants will receive single dose of LY3009104 on 4 separate occasions with and without food. Safety evaluation and serial pharmacokinetic (PK) samples will be collected during each treatment period. Approximately 5 to 7 days of washout period between each treatment and a follow-up visit will occur approximately 5 to 7 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females as determined by medical history and physical examination
* Have a body mass index (BMI) of 18.5 to 29.9 kilograms per square meter (kg/m^2), inclusive, at screening
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have normal blood pressure and pulse rate as determined by the investigator
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Male Participants:

* Agree to use two forms of highly effective methods of birth control [oral, injectable, or implanted hormonal contraceptives; condom with spermicidal foam/gel/film/cream/suppository; occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; intrauterine device; intrauterine system, for example, progestin releasing coil; and vasectomised male (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate)] with female partners of childbearing potential during the study and for at least 3 months following the last dose of study drug

Female participants:

* Are women of non-childbearing potential, defined as: women with Mayer Rokitansky Kuster Hauser Syndrome (also referred to as Clinical Absence of Uterus and Vagina), or women who have had surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation), or women greater than 60 years of age, or women greater than 40 and less than 60 years of age who have had a cessation of menses for at least 12 months and a follicle-stimulating hormone (FSH) test confirming non-childbearing potential [FSH ≥40 milli-international units per milliliter (mIU/mL)]

Exclusion Criteria:

* Are currently enrolled in, or have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have a history of adverse drug reactions or "drug allergy" to more than 3 types of systemically administered medications (all penicillins and cephalosporins may be considered 1 type of medication for this purpose)
* Are participants who have previously received the investigational product in this study, have completed or withdrawn from this study or any other study investigating LY3009104
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Current or recent history (<30 days prior to screening and/or <45 days prior to Check-in) of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
* Have an absolute neutrophil count (ANC) less than 2000 cells per microliter (cell/μL). For abnormal values, a single repeat will be allowed
* Have a history of, or current, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Regularly use known drugs of abuse
* Have had symptomatic herpes zoster or herpes simplex infection within 90 days prior to the first dose
* Have been exposed to a live vaccine within 12 weeks prior to the first dose or expected to need/receive a live vaccine (including herpes zoster vaccination) during the course of the study
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Intend to use over-the-counter or prescription medication and herbal supplements within 14 days prior to dosing and during the study
* Intend to use vitamins and mineral supplements within 2 days prior to dosing and during the study
* Have donated blood of more than 450 milliliters (mL) within the previous 3 months
* Have consumed grapefruit, starfruit, pomelos, or products containing these fruits, 7 days prior to the first dose and during the study
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to stop alcohol consumption for 48 hours prior to admission in each period until the 48 hour PK sample has been collected [1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Have used any tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- LY3009104 (LY) RF, LY 50-mcm Fed, LY 20-mcm, LY 50-mcm Fasted: First intervention: 8-milligram (mg) dose of LY3009104 reference formulation (RF, two 4-mg phosphate salt capsules) administered once in a fasted state.
  Second intervention: 8-mg dose of LY3009104 test formulation 2 [TF2, one 8-mg tablet, free base formulation, target active pharmaceutical ingredient (API) particle size of 50 micrometers (mcm)] administered once with a high-fat, high calorie meal.
  Third intervention: 8-mg dose of LY3009104 test formulation 1 (TF1, one 8-mg tablet, free base formulation, target API particle size of 20 mcm) administered once in a fasted state.
  Fourth intervention: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once in a fasted state.
  There was a washout period of 5 to 7 days between doses of study drug.
- LY 20-mcm, LY RF, LY 50-mcm Fasted, LY 50-mcm Fed: First intervention: 8-mg dose of LY3009104 TF1 (one 8-mg tablet, free base formulation, target API particle size of 20 mcm) administered once in a fasted state.
  Second intervention: 8-mg dose of LY3009104 RF (two 4-mg phosphate salt capsules) administered once in a fasted state.
  Third intervention: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once in a fasted state.
  Fourth intervention: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once with a high-fat, high calorie meal.
  There was a washout period of 5 to 7 days between doses of study drug.
- LY 50-mcm Fasted, LY 20-mcm, LY 50-mcm Fed, LY RF: First intervention: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once in a fasted state.
  Second intervention: 8-mg dose of LY3009104 TF1 (one 8-mg tablet, free base formulation, target API particle size of 20 mcm) administered once in a fasted state.
  Third intervention: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once with a high-fat, high calorie meal.
  Fourth intervention: 8-mg dose of LY3009104 RF (two 4-mg phosphate salt capsules) administered once in a fasted state.
  There was a washout period of 5 to 7 days between doses of study drug.
- LY 50-mcm Fed, LY 50-mcm Fasted, LY RF, LY 20-mcm: First intervention: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once with a high-fat, high calorie meal.
  Second intervention: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once in a fasted state.
  Third intervention: 8-mg dose of LY3009104 RF (two 4-mg phosphate salt capsules) administered once in a fasted state.
  Fourth Intervention: 8-mg dose of LY3009104 TF1 (one 8-mg tablet, free base formulation, target API particle size of 20 mcm) administered once in a fasted state.
  There was a washout period of 5 to 7 days between doses of study drug.
Period: Overall Study
Arm/Group | LY3009104 (LY) RF, LY 50-mcm Fed, LY 20-mcm, LY 50-mcm Fasted | LY 20-mcm, LY RF, LY 50-mcm Fasted, LY 50-mcm Fed | LY 50-mcm Fasted, LY 20-mcm, LY 50-mcm Fed, LY RF | LY 50-mcm Fed, LY 50-mcm Fasted, LY RF, LY 20-mcm
Started | 4 | 3 | 4 | 4
Received First Intervention | 4 | 3 | 4 | 4
Received Second Intervention | 4 | 3 | 4 | 4
Received Third Intervention | 4 | 3 | 4 | 4
Received Fourth Intervention | 4 | 3 | 4 | 4
Completed | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Entire Study Population: Includes groups randomized to receive any of the following study drugs as the first intervention.
  LY3009104 Reference Formulation (RF): 8-milligram (mg) dose of LY3009104 RF (two 4-mg phosphate salt capsules) administered once in a fasted state.
  LY3009104 Test Formulation 1 (TF1), 20 micrometers (mcm): 8-mg dose of LY3009104 TF1 [one 8-mg tablet, free base formulation, target active pharmaceutical ingredient (API) particle size of 20 mcm] administered once in a fasted state.
  LY3009104 Test Formulation 2 (TF2), 50 mcm, fasted: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once in a fasted state.
  LY3009104 TF2, 50 mcm, fed: 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once with a high-fat, high calorie meal.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 14
  White | 1
Region of Enrollment [Number; unit: participants]
  Singapore | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Plasma Concentration-Time Curve (AUC)
Description: The area under the concentration-time curve from time 0 to infinity [AUC(0-inf)] is reported for participants who received either LY3009104 tablets or capsules in a fasted or fed state.
Time Frame: Predose up to 48 hours postdose for each of the 4 treatment periods
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hours per liter (nmol*h/L)
Groups:
- LY3009104 Reference Formulation: 8-milligram (mg) dose of LY3009104 reference formulation (RF, two 4-mg phosphate salt capsules) administered once in a fasted state in Period 1, 2, 3, or 4.
- LY3009104 Test Formulation 1 (20-mcm): 8-mg dose of LY3009104 test formulation 1 [TF1, one 8-mg tablet, free base formulation, target active pharmaceutical ingredient (API) particle size of 20 micrometers (mcm)] administered once in a fasted state in Period 1, 2, 3, or 4.
- LY3009104 Test Formulation 2 (50-mcm, Fed): 8-mg dose of LY3009104 test formulation 2 (TF2, one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once with a high-fat, high calorie meal in Period 1, 2, 3, or 4.
- LY3009104 Test Formulation 2 (50-mcm, Fasted): 8-mg dose of LY3009104 TF2 (one 8-mg tablet, free base formulation, target API particle size of 50 mcm) administered once in a fasted state in Period 1, 2, 3, or 4.
Arm/Group | LY3009104 Reference Formulation | LY3009104 Test Formulation 1 (20-mcm) | LY3009104 Test Formulation 2 (50-mcm, Fed) | LY3009104 Test Formulation 2 (50-mcm, Fasted)
Number analyzed (Participants) | 15 | 15 | 15 | 15
nanomoles*hours per liter (nmol*h/L) | 1670 (35) | 1710 (32) | 1510 (34) | 1700 (35)
Statistical Analysis 1: Comparison: LY3009104 Reference Formulation vs LY3009104 Test Formulation 1 (20-mcm); Test type: Superiority or Other; Geometric least squares (LS) mean ratio = 1.02, 90% CI 2-sided [0.951 to 1.10] — The geometric LS mean ratio (TF1 fasted divided by RF fasted) was calculated using a linear mixed-effects model adjusted for treatment, sequence, period, and participant
Statistical Analysis 2: Comparison: LY3009104 Reference Formulation vs LY3009104 Test Formulation 2 (50-mcm, Fasted); Test type: Superiority or Other; Geometric LS mean ratio = 1.02, 90% CI 2-sided [0.947 to 1.09] — The geometric LS mean ratio (TF2 fasted divided by RF fasted) was calculated using a linear mixed-effects model adjusted for treatment, sequence, period, and participant
Statistical Analysis 3: Comparison: LY3009104 Test Formulation 2 (50-mcm, Fed) vs LY3009104 Test Formulation 2 (50-mcm, Fasted); Test type: Superiority or Other; Geometric LS mean ratio = 0.888, 90% CI 2-sided [0.827 to 0.953] — The geometric LS mean ratio (TF2 fed divided by TF2 fasted) was calculated using a linear mixed-effects model adjusted for treatment, sequence, period, and participant

2. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax)
Time Frame: Predose up to 48 hours postdose for each of the 4 treatment periods
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Arm/Group | LY3009104 Reference Formulation | LY3009104 Test Formulation 1 (20-mcm) | LY3009104 Test Formulation 2 (50-mcm, Fed) | LY3009104 Test Formulation 2 (50-mcm, Fasted)
Number analyzed (Participants) | 15 | 15 | 15 | 15
nanomoles per liter (nmol/L) | 259 (26) [231 to 286] | 253 (19) [226 to 280] | 205 (27) | 250 (30) [222 to 275]
Statistical Analysis 1: Comparison: LY3009104 Reference Formulation vs LY3009104 Test Formulation 1 (20-mcm); Test type: Superiority or Other; Geometric least squares (LS) mean ratio = 0.979, 90% CI 2-sided [0.868 to 1.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: LY3009104 Reference Formulation vs LY3009104 Test Formulation 2 (50-mcm, Fasted); Test type: Superiority or Other; Geometric LS mean ratio = 0.962, 90% CI 2-sided [0.852 to 1.08] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: LY3009104 Test Formulation 2 (50-mcm, Fed) vs LY3009104 Test Formulation 2 (50-mcm, Fasted); Test type: Superiority or Other; Geometric LS mean ratio = 0.820, 90% CI 2-sided [0.727 to 0.925] — [estimate comment as in outcome 1, analysis 3]

3. Secondary Outcome: Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax)
Time Frame: Predose up to 48 hours postdose for each of the 4 treatment periods
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | LY3009104 Reference Formulation | LY3009104 Test Formulation 1 (20-mcm) | LY3009104 Test Formulation 2 (50-mcm, Fed) | LY3009104 Test Formulation 2 (50-mcm, Fasted)
Number analyzed (Participants) | 15 | 15 | 15 | 15
hours (h) | 1.00 [0.50 to 3.00] | 1.00 [0.50 to 3.00] | 2.00 [1.00 to 4.00] | 1.00 [0.50 to 2.00]
Statistical Analysis 1: Comparison: LY3009104 Reference Formulation vs LY3009104 Test Formulation 1 (20-mcm); Test type: Superiority or Other; p = 0.719, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 90% CI 2-sided [-0.250 to 0.500] — The median difference was calculated as TF1 fasted minus RF fasted
Statistical Analysis 2: Comparison: LY3009104 Reference Formulation vs LY3009104 Test Formulation 2 (50-mcm, Fasted); Test type: Superiority or Other; p = 0.960, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 90% CI 2-sided [-0.250 to 0.750] — The median difference was calculated as TF2 fasted minus RF fasted
Statistical Analysis 3: Comparison: LY3009104 Test Formulation 2 (50-mcm, Fed) vs LY3009104 Test Formulation 2 (50-mcm, Fasted); Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.500, 90% CI 2-sided [0 to 2.00] — The median difference was calculated as TF2 fed minus TF2 fasted

ADVERSE EVENTS:
Groups:
- LY3009104 Test Formulation 2 (50-mcm, Fed): 8-mg dose of LY3009104 test formulation 2 [TF2, one 8-mg tablet, free base formulation, target active pharmaceutical ingredient (API) particle size of 50 micrometer (mcm)] administered once with a high-fat, high calorie meal in Period 1, 2, 3, or 4.
- LY3009104 Test Formulation 1 (20-mcm): 8-mg dose of LY3009104 test formulation 1 (TF1, one 8-mg tablet, free base formulation, target API particle size of 20 mcm) administered once in a fasted state in Period 1, 2, 3, or 4.
Arm/Group | LY3009104 Reference Formulation | LY3009104 Test Formulation 2 (50-mcm, Fed) | LY3009104 Test Formulation 1 (20-mcm) | LY3009104 Test Formulation 2 (50-mcm, Fasted)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 5/15 | 2/15 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3009104 Reference Formulation (N=15) | LY3009104 Test Formulation 2 (50-mcm, Fed) (N=15) | LY3009104 Test Formulation 1 (20-mcm) (N=15) | LY3009104 Test Formulation 2 (50-mcm, Fasted) (N=15)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes